CLINICAL TRIAL: NCT03527134
Title: Effects of Amantadine on Postoperative Cognitive Dysfunction in Elderly Patients With Elective Abdominal Surgery
Brief Title: Effects of Amantadine on Postoperative Cognitive Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhiyi Zuo (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Zhiyi Zuo, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-34
Record Dates: First submitted 2018-04-23; First posted 2018-05-17 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Amantadine

STUDY DESIGN:
Intervention Model Description: Two groups: one with amantadine treatment and the other with amantadine treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amantadine treatment (Experimental): To determine whether amantadine is effective in reducing the occurrence of postoperative cognitive dysfunction.
  Interventions: Drug: Amantadine
- No-treatment (No Intervention): Patients will not receive any treatment.

INTERVENTIONS:
Drug: Amantadine — patients will receive amantadine 100 mg by month 2 h before the induction of general anesthesia and then 100 mg each time, three times per day for 5 days.
  Arms: Amantadine treatment

SUMMARY:
Post-operative cognitive dysfunction (POCD) is a fairly well-documented clinical phenomenon. Investigators will determine whether amantadine can reduce the occurrence of POCD in elderly patients with major abdominal surgery.

DETAILED DESCRIPTION:
Patients who are 60 years old or older for laparoscopic abdominal surgery will be randomly assigned into two groups: 1) no-treatment group, and 2) amantadine-treated group. Each group will have 150 patients. In addition, investigators will need 90 subjects in the control group. The data of these control subjects will be used to normalize the data of the two studied groups to diagnose POCD. The subjects in control groups will also be elderly but without the exposure to anesthesia and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. major elective gynecological, prostate or bladder surgery patients who are ≥ 60 years old.
2. the surgery is laparoscopic surgery and is expected to last for ≥ 2 hours under general anesthesia and the patient will stay in hospital for at least 7 days after surgery.
3. lack of serious hearing and vision impairment and be able to read so that neurobehavioral tests can be performed.

Exclusion Criteria:

1. Patients are not expected to be alive for longer than 3 months.
2. Mini-mental State Examination (MMSE) [18] score ≤ 23.
3. history of dementia, psychiatric illness or any diseases of central nervous system.
4. current use of sedatives or antidepressant.
5. alcoholism and drug dependence.
6. patients previously included in this study (for patients who have second intra-abdominal surgery during the study period).
7. difficult to follow up or patients with poor compliance.
8. uncontrolled hypertension (> 180/100 mmHg)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction (POCD) (POCD is a composite outcome measure) | At 7 days after the surgery
  The existence of POCD will be determined by Visual Verbal Learning Test based on the Rey's Auditory Recall of words, Concept Shifting Test, Stroop Color Word Interference Test and Letter-Digit Coding based on the Symbol Digit Substitution Test

SECONDARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction (POCD) (POCD is a composite outcome measure) | At 3 months after the surgery
  The existence of POCD will be determined by Visual Verbal Learning Test based on the Rey's Auditory Recall of words, Concept Shifting Test, Stroop Color Word Interference Test and Letter-Digit Coding based on the Symbol Digit Substitution Test
Time for bowel function return after surgery | up to 2 weeks after the surgery
Degree of increase of stress hormone | Up to 5 days after the surgery
  Adrenocorticotropic Hormone
Length of hospital stay | Up to 3 months after the surgery
Degree of change in growth factor | Up to 5 days after the surgery
  Brain-derived neurotrophic factor and glial cell derived neurotrophic factor

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China